CLINICAL TRIAL: NCT04235855
Title: EUS Guided Liver Biopsy Proposal Titled : EUS Guided Liver Biopsy - Will it Give Better Yield , More Tissue With Less Complication ?
Brief Title: EUS Guided Liver Biopsy - Will it Give Better Yield, More Tissue With Less Complication?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Dr Mithun Sharma, Consultant Hepatologist, Asian Institute of Gastroenterology, India
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ECR/346/Inst/AP/2013/RR-19
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: NAFLD; Alcoholic Hepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hepatitis, Alcoholic

STUDY DESIGN:
Intervention Model Description: All liver biopsies done in the Institute as routine procedure by percutaneous route would be compared with the EUS guided biopsy in respect to safety , tissue quality and diagnostic yield.
Who Masked: Outcomes Assessor
Masking Description: The biopsy specimens would be reported independently by two pathologists who would be masked to the source of tissue ( right/ left lobe ).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic USG guided Liver biopsy (Experimental): Olympus linear echo endoscope (GF -UCT 180, Olympus Ltde, Tkyo, Japan) will be used. 19 Gz EUS Acquire needle Boston ©Scientific Corp will be used for liver tissue acquisition.
  Interventions: Device: Endoscopic USG guided Liver biopsy
- Percutaneous Liver biopsy (Active Comparator): All liver biopsies done in the Institute as routine procedure by percutaneous route would be compared with the EUS guided biopsy in respect to safety , tissue quality and diagnostic yield .
  Interventions: Device: Percutaneous Liver Biopsy

INTERVENTIONS:
Device: Endoscopic USG guided Liver biopsy — Diagnostic yield with EUS guided liver biopsy - Left lobe Bx vs combined right and left lobe or vs right lobe would be assessed.
  Arms: Endoscopic USG guided Liver biopsy
Device: Percutaneous Liver Biopsy — All liver biopsies done in the Institute as routine procedure by percutaneous route would be compared with the EUS guided biopsy in respect to safety , tissue quality and diagnostic yield .
  Arms: Percutaneous Liver biopsy

SUMMARY:
Liver biopsy would be done by Endoscopic Ultrasound using Acquire needle.

DETAILED DESCRIPTION:
In this study, we aim to evaluate the tissue adequacy of EUS guided liver biopsy for parenchymal liver disease and to evaluate if diagnostic yield of left lobe is non-inferior to right lobe biopsies and to assess if combination biopsies have better yield than single lobe biopsies. Safety of the procedure and technical success would be noted.

The data would be analysed using SPSS software and needful variables and tests would be used as per statistical requirement.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any undiagnosed hepatic disease (after extensive investigation - serological as well as imaging) requiring a liver biopsy
* Patients of NAFLD who need liver biopsy
* Alcoholic hepatitis patients needing biopsy
* Any patient with unexplained transaminesemia > 1.5 times ULN needing a liver biopsy as advised by Hepatologist

Exclusion Criteria:

* Any liver Space occupying lesion suspicious of malignancy
* Platelet count <80,000
* INR > 1.5
* Pregnancy
* Severe cardiovascular and pulmonary diseases
* Recent use of anti-platelet agents within 5 days of the procedure
* Unwilling to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield with EUS guided liver biopsy . | 3 days
  The diagnostic yield of a right lobe biopsy and left lobe biopsy would be compared to see if right lobe biopsy gives any additional information for diagnosis when compared to left lobe .

SECONDARY OUTCOMES:
Safety of procedure | 3 days
  Sedation related adverse effect will be monitored as per the institute protocol . Any type of bleed during procedure or needing additional intervention would be recorded as a major adverse effect .
Duration of procedure | 30 minutes
  Time between start and end of the procedure would be noted .
Size of tissue acquired | 3 days
  The length of the biopsy tissue would be ascertained immediately by onsite pathologist and would be assessed as per the AASLD and Royal College of Pathology definition .
Number of portal tracts | 3 days
  The adequacy of the sample would be assessed as per the AASLD and Royal College of Pathology definition (CPTs 11) .
Post procedural complications | 3 days
  Any procedure related complications such as pain (>6 on VAS) and bleeding would be noted .
NAS score in fatty liver patients | 3 days
  Difference in NAS score between right lobe and right vs left lobe in fatty liver patients
Patient recovery time | 3 days
  Patient recovery time when compared to per cutaneous liver biopsy procedure .

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology Hospitals, Hyderabad, Telangana, India

REFERENCES:
- [Background] Gor N, Salem SB, Jakate S, Patel R, Shah N, Patil A. Histological adequacy of EUS-guided liver biopsy when using a 19-gauge non-Tru-Cut FNA needle. Gastrointest Endosc. 2014 Jan;79(1):170-2. doi: 10.1016/j.gie.2013.06.031. Epub 2013 Jul 31. No abstract available. PMID 23916397
- [Background] Dewitt J, McGreevy K, Cummings O, Sherman S, Leblanc JK, McHenry L, Al-Haddad M, Chalasani N. Initial experience with EUS-guided Tru-cut biopsy of benign liver disease. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):535-42. doi: 10.1016/j.gie.2008.09.056. PMID 19231495
- [Background] Schulman AR, Thompson CC, Odze R, Chan WW, Ryou M. Optimizing EUS-guided liver biopsy sampling: comprehensive assessment of needle types and tissue acquisition techniques. Gastrointest Endosc. 2017 Feb;85(2):419-426. doi: 10.1016/j.gie.2016.07.065. Epub 2016 Aug 13. PMID 27530070